CLINICAL TRIAL: NCT06976632
Title: Comparison of the Effects of the Helfer Skin Tap Technique and Local Cold Application on Pain and Hemodynamic Parameters During Vaccination in Pregnant Women
Brief Title: Effect of Helfer Skin Tap and Cold Application on Pain and Hemodynamics During Vaccination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Sevgi Çetin, Asst. Prof., Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20.478.486/2967
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pregnant Women
Keywords: immunization; pain; hemodynamic parameters; pregnant women; local cold application; helfer skin tap tecnique
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The pregnant women to be assigned to the group will be determined using the Research Randomizer program. In the first phase of the study, pregnant women who accept to participate and meet the sample selection criteria will be informed about the study, and written and verbal consent will be obtained. Then, before the intramuscular tetanus vaccination, a "Personal Information Form" will be filled out by one of the researchers, the institution nurse, using a face-to-face interview technique. In the second phase, the nurse will measure the vital signs of the pregnant women. Then, the vaccine will be administered using the method used. In the third phase of the study, pain assessment will be made using the NPS immediately after the procedure and 15 minutes later, and the vital signs of the pregnant women will be measured. Pain evaluation will be conducted 24 and 48 hours after the vaccination.
Who Masked: Participant
Masking Description: In this study, participants were randomly assigned to groups in order to evaluate the effectiveness of nursing interventions. Randomization was carried out by creating 3 sets, each containing 30 unique numbers ranging from 1 to 90. Each set was used for group assignments. The randomization process was organized sequentially with non-repeating numbers across the sets. Participants were assigned to groups according to the order of each set. The randomization process was performed using the Research Randomizer program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The injection is administered using the standard method.
- Helfer Skin Tap Tecnique (Experimental): After identifying the injection site, the muscles are relaxed by gently tapping the skin with the fingertips of the dominant hand for about five seconds. Using the thumb and index finger of the non-dominant hand, a V shape is formed, and the entire hand is used to tap the skin three times. Simultaneously with the third tap, the needle is inserted into the muscle at a 90-degree angle. After aspiration, the medication is injected over 5 seconds while continuing to gently tap the skin with the fingertips of the non-dominant hand. After administering the medication, the needle is withdrawn from the muscle simultaneously with final tap, while tapping the skin in a V shape using the non-dominant hand.
  Interventions: Behavioral: Helfer Skin Tap Tecnique
- Local Cold Application (Experimental): A cold gel compress is removed from the freezer and left at room temperature for a few minutes to thaw slightly. After identifying the injection site, the cold gel compress is wrapped in gauze and placed on the deltoid area to cover the injection site. The cold gel compress is held in place for one minute. After one minute, the cold gel compress is removed. The skin is cleaned with an alcohol swab, then the injection is administered.
  Interventions: Behavioral: Local Cold Application

INTERVENTIONS:
Behavioral: Helfer Skin Tap Tecnique — In the first phase of the study, pregnant women who agree to participate and meet the sampling criteria will be informed about the study, and their written and verbal consents will be obtained. Then, the "Individual Identification Form" will be completed.
  In the second phase, the vital signs of the pregnant women will be measured by the nurse involved in the study. Following this, tetanus vaccination will be administered to the pregnant women in the intervention group using the Helfer Skin Tap technique in accordance with the "Helfer Skin Tap IM Injection Procedure Guideline".
  In the third phase of the study, pain will be assessed using the Numerical Pain Scale immediately after the procedure and 15 minutes later by the nurse, and the vital signs of the pregnant women will be measured again. To evaluate the long-term effects of pain, participants will be contacted via a link, and pain assessments will be conducted at the 24th and 48th hours following the vaccination.
  Arms: Helfer Skin Tap Tecnique
Behavioral: Local Cold Application — In the first phase of the study, pregnant women who agree to participate and meet the sampling criteria will be informed about the study, and their written and verbal consents will be obtained. Then, the "Individual Identification Form" will be completed.
  In the second phase, the vital signs of the pregnant women will be measured by the nurse involved in the study. Subsequently, tetanus vaccination will be administered to the pregnant women in the intervention group using a cold compress gel, based on the "Cold Compress Gel IM Injection Procedure Guideline" developed in line with the relevant literature.
  In the third phase of the study, pain will be assessed using the Numerical Pain Scale immediately after the procedure and 15 minutes later by nurse, and the vital signs of the pregnant women will be measured again. Pain assessment will be repeated at the 24th and 48th hours following the vaccination.
  Arms: Local Cold Application

SUMMARY:
The purpose of this study is to investigate the effect of local cold application using the Helfer Skin Tap Technique on pain levels during the intramuscular injection of the tetanus vaccine in pregnant women. The study will also record vital signs, which are among the physiological effects of pain.

DETAILED DESCRIPTION:
This randomized controlled study aims to evaluate the effects of the Helfer Skin Tap Technique and local cold application on pain intensity and hemodynamic parameters during intramuscular tetanus vaccination in pregnant women. The sample size will be calculated prior to data collection using the G*Power 3.1.9.2 software. Pregnant women included in the sample will be randomly assigned to three groups using the Research Randomizer program.

According to the randomization:

Group 1 (intervention) will receive the tetanus vaccine using the Helfer Skin Tap Technique, Group 2 (intervention) will receive the vaccine with local cold application, Group 3 (control) will receive the standard IM injection without additional intervention.

Data will be collected from pregnant women who are followed by Soma No. 5 Family Health Center and who apply to the institution for tetanus vaccination during pregnancy. The data collection tools include a Personal Information Form, Numeric Pain Rating Scale (NPRS), the Helfer Skin Tap IM Injection Procedure Guideline, Cold Compress Gel IM Injection Guideline, and Standard IM Injection Guideline.

Injections will be administered to participants in all groups according to the respective guidelines. Vital signs (such as heart rate, blood pressure, peripheral oxygen saturation (%), and respiratory rate) will be measured before injection, immediately after injection, and 15 minutes post-injection. Pain levels will be assessed immediately and at the 15th minute following the injection. Additionally, to evaluate the longer-term effects of pain, participants will be contacted via a follow-up link and asked to report their pain levels at the 24th and 48th hours after vaccination.

ELIGIBILITY:
Inclusion Criteria: Pregnant women who meet the following criteria will be included in the study:

* Over the age of 18,
* Scheduled to receive a tetanus vaccine,
* Able to speak and communicate in Turkish,
* Willing to participate in the study,
* Not experiencing any pain for any reason prior to the injection.

Exclusion Criteria: Pregnant women who meet any of the following criteria will be excluded from the study:

* Under the age of 18,
* Received a tetanus vaccine for reasons other than pregnancy,
* Received a vaccine other than tetanus,
* Experiencing pain for any reason prior to the vaccine,
* Have circulatory disorders or peripheral vascular disease,
* Have bleeding or clotting disorders,
* Have a local infection,
* Used painkillers at least 6 hours prior to the procedure,
* Underwent a painful procedure within the last hour,
* Have cold sensitivity,
* Have cognitive or psychological issues.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Individuals over the age of 18 who have received the tetanus vaccine due to pregnancy.
Enrollment: 90 (Estimated)
Dates: Start 2025-05-09 (Estimated); Primary Completion 2026-05-09 (Estimated); Study Completion 2026-05-09 (Estimated)

PRIMARY OUTCOMES:
Individual Identification Form | It was implemented on the first day of the study.
  The "Individual Identification Form," which includes the sociodemographic characteristics of the pregnant women, was developed by the researchers based on the relevant literature. The form consists of 9 questions.
Use of a numerical pain scale in the assessment of injection-related pain | immediately after the injection, 15 minutes later, and at the 24th and 48th hours
  Pain assessment related to the injection in pregnant women will be conducted using the Numerical Pain Scale immediately after the injection, 15 minutes later, and at the 24th and 48th hours. It is based on the principle that patients circle the number representing the amount of pain they experience on a 10 cm horizontal scale, with "No Pain" written at the far left and "Severe Pain" at the far right. When evaluating pain intensity, a score of 0 indicates "No pain," 1-3 points indicate "Mild pain," 4-6 points indicate "Moderate pain," and 7-10 points indicate "Severe pain."

SECONDARY OUTCOMES:
Monitoring the systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg) of the pregnant women | before the injection, immediately after the injection, and 15 minutes after the injection
  In the study, systolic blood pressure (mm/Hg) and diastolic blood pressure (mm/Hg), which is one of the physiological effects of pain, will be recorded three times.
Monitoring the heart rate (per minute) of the pregnant women | before the injection, immediately after the injection, and 15 minutes after the injection
  In the study, heart rate (per minute), which is one of the physiological effects of pain, will be recorded three times.
Monitoring the respiratory rate (per minute) of the pregnant women | before the injection, immediately after the injection, and 15 minutes after the injection
  In the study, respiratory rate (per minute), which is one of the physiological effects of pain, will be recorded three times.
Monitoring the peripheral oxygen saturation (%) of the pregnant women | before the injection, immediately after the injection, and 15 minutes after the injection
  In the study, peripheral oxygen saturation (%), which is one of the physiological effects of pain, will be recorded three times.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Pakiş Çetin, Asst. Prof., Principal Investigator — Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Manisa, Uncubozköy/Yunusemre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It can be shared upon request, if the relevant ethics committee approves.
Supporting Information: CSR
Time Frame: Starting 6 months after publication.
Access Criteria: It can be shared upon request, if the relevant ethics committee approves.